CLINICAL TRIAL: NCT03644004
Title: Descriptive Study of the Diabetes Mellitus, Type 2 Diagnosis Methods During Postpartum Period in Patients With Medical History of Gestational Diabetes Whom Benefited an Educational Therapy Session.
Brief Title: Oral Glucose Tolerance Test and Post Partum Diagnosis of Diabetes Mellitus, Type 2 (DT2 Post-Partum)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0210
Record Dates: First submitted 2018-08-16; First posted 2018-08-23 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with medical history of gestational diabetes: Patients followed at the hospital of Vienne for gestational diabetes in 2016.
  Interventions: Other: frequency of diabetes mellitus, type 2, diagnosis in patients with medical history of gestational diabetes.

INTERVENTIONS:
Other: frequency of diabetes mellitus, type 2, diagnosis in patients with medical history of gestational diabetes. — Patients will be contacted by mail with sending of the information notice to ask them to participate in the study.
  If they don't reply, the subjects will be called by phone by the investigator to collect their non opposition of participation at the study.
  During this call, the investigator will be able to answer all the questions about the study.
  The report of this telephone conversation will be register in the medical file of the patient.
  Then, we will collect informatic data from the hospital concerning the patients.
  After that they will be contacted by phone to answer a survey. Beside, another secure survey will be send by email to each patient's family doctor.
  To finish, crossing data between those of the patients and the family doctor and anonymisation of the data.
  Other Names: Evaluate the frequency of diabetes mellitus, type 2, diagnosis with an oral glucose tolerance test between 6 and 12 weeks after childbirth in patients with medical history of gestational diabetes.

SUMMARY:
Diabetes mellitus, type 2, is a chronic disease which can be linked with many complications in connexion with impaired blood glucose balance.

It diagnosis in risky subjects such as in patients with medical history of gestational diabetes is therefore imperative to prevent its complications.

Actual guidelines recommend an oral tolerance glucose test, measuring glucose levels after oral glucose intake (75g), between 6 an 12 weeks after childbirth. But studies reveal a low diagnosis rate.

The study of the current practices of diagnosis methods seem to be essential in order to improve this diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in endocrinology at the hospital of Vienne for gestational diabetes, whom benefited an educational therapy session between the 01/01/2016 and the 31/12/2016 inclusive.

Exclusion Criteria:

* Minor patients or under legal protection (guardianship)
* Patients who not speak french
* Patients who did not declared an attending physician
* Refusal to take part in the survey
* Patients lost to follow-up before childbirth
* Patients whose pregnancy ended by foetal death.
* Pre-existing diabet before pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who develop a gestational diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Performing oral glucose tolerance test in order to detect type 2 diabetes | Month 6
  Performing oral glucose tolerance test between 6 and 12 weeks after childbirth. As recommended by actual World Health Organisation (WHO) guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Laura BOGENMANN, MD, Study Director — Centre Hospitalier de Vienne
Locations (1):
- Centre hospitalier Lucien Hussel, Vienne, France